CLINICAL TRIAL: NCT07053527
Title: Welcome to PrEP School Utilizing Peer Educators to Improve Uptake of Preexposure Prophylaxis for HIV at an HBCU
Acronym: PrEPSchool
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Morehouse School of Medicine (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Principal Investigator, Kara Garretson, MPH, Sr. Epidemiologist and Infection, Prevention & Control Safety Officer for AUCC Student Health Division, Morehouse School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2264597
Record Dates: First submitted 2025-06-02; First posted 2025-07-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-05

CONDITIONS: HIV Prevention Program
Keywords: Preexposure Prophylaxis; PrEP Awareness; PrEP Access; PrEP Uptake; HIV Prevention; Peer education; HBCU

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Educational Intervention Arm: African American College Students Receiving PrEP Awareness Sessions (Experimental): Develop a peer-educator/navigation intervention to help decrease stigma and discrimination and foster knowledge around PrEP use, in the prevention of HIV
  Interventions: Behavioral: PrEP Awareness and Uptake Educational Program

INTERVENTIONS:
Behavioral: PrEP Awareness and Uptake Educational Program — This intervention targets African American college students aged 18-26 using a tailored, community participatory approach. It is delivered by trained peer educators and focuses on increasing PrEP awareness, access, and uptake through interactive, behaviorally focused sessions. Developed with input from focus groups to ensure relevance, the program includes a 6-month follow-up to assess sustained impact, distinguishing it from general PrEP education efforts.

SUMMARY:
This study involves a peer-educator/navigation model targeting gaps in PrEP awareness, uptake, and access in priority populations.

DETAILED DESCRIPTION:
The study focuses on increasing awareness and uptake of Pre-Exposure Prophylaxis (PrEP) for HIV prevention among African American college students at a consortium of historically Black colleges and universities in Atlanta, GA.

ELIGIBILITY:
Inclusion Criteria:

* 18-26 years old
* not currently on PrEP
* English speaking
* HIV negative
* 5) Enrolled in the following universities: Spellman College, Morehouse College, Clark Atlanta University, Morehouse school of medicine

Exclusion Criteria:

* Age < 18 years old
* Non-English speaking
* HIV positive
* Not currently enrolled any of the four colleges/universities

Ages: 18 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 123 (Estimated)
Dates: Start 2025-06-28 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Welcome to PrEP School Utilizing Peer Educators to Improve Uptake of Pre-Exposure Prophylaxis for HIV at an HBCU Consortium | 12 months
  The Primary endpoint will be increased awareness, acceptability and access of PrEP by measuring pre-post surveys after peer-educator/navigator educational intervention.

SECONDARY OUTCOMES:
Welcome to PrEP School Utilizing Peer Educators to Improve Uptake of Pre-Exposure Prophylaxis for HIV at an HBCU Consortium | 12 months
  The secondary endpoint will be measuring clinic data assessing the proportion of college students who initiated PrEP post educational intervention over a 12 months period.

CONTACTS AND LOCATIONS:
Overall Officials: Kara Garretson, Principal Investigator — Morehouse School of Medicine
Locations (1):
- Morehouse School of Medicine, Atlanta, Georgia, United States

REFERENCES:
- [Background] Weber S, Lazar L, McCord A, Romero C, Tan J. Online Navigation for Pre-Exposure Prophylaxis via PleasePrEPMe Chat for HIV Prevention: Protocol for a Development and Use Study. JMIR Res Protoc. 2020 Sep 22;9(9):e20187. doi: 10.2196/20187. PMID 32960183
- [Background] Truong HM, Pipkin S, O'Keefe KJ, Louie B, Liegler T, McFarland W, Grant RM, Bernstein K, Scheer S. Brief Report: Recent Infection, Sexually Transmitted Infections, and Transmission Clusters Frequently Observed Among Persons Newly Diagnosed With HIV in San Francisco. J Acquir Immune Defic Syndr. 2015 Aug 15;69(5):606-9. doi: 10.1097/QAI.0000000000000681. PMID 25967271
- [Background] Pichon LC, Teti M, McGoy S, Murry VM, Juarez PD. Engaging Black men who have sex with men (MSM) in the South in identifying strategies to increase PrEP uptake. BMC Health Serv Res. 2022 Dec 7;22(1):1491. doi: 10.1186/s12913-022-08914-2. PMID 36476363
- [Background] Okeke NL, McLaurin T, Gilliam-Phillips R, Wagner DH, Barnwell VJ, Johnson YM, James O, Webb PB, Parker SD, Hill B, McKellar MS, Mitchell JT. Awareness and acceptability of HIV pre-exposure prophylaxis (PrEP) among students at two historically Black universities (HBCU): a cross-sectional survey. BMC Public Health. 2021 May 19;21(1):943. doi: 10.1186/s12889-021-10996-2. PMID 34006245